CLINICAL TRIAL: NCT03810950
Title: Physiological, Neural and Behavioral Correlates of Psychosocial Stress and Alcohol Craving
Brief Title: Psychobiology of Stress and Alcohol Craving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Project Group for Automation in Medicine and Biotechnology PAMB, Mannheim (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 A03-Pilot
Record Dates: First submitted 2018-11-26; First posted 2019-01-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Alcohol Use Disorder; Stress Reaction; Social Stress; Craving; Behavior
MeSH Terms: conditions — Alcoholism; Fractures, Stress; Behavior | interventions — Psychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Stress Test (Experimental): Participants undergo the Trier Social Stress Test before Barlab-Exposure
  Interventions: Behavioral: Trier Social Stress Test; Behavioral: Barlab-Exposure
- Control Condition (Active Comparator): Participants reads newspaper before Barlab-Exposure
  Interventions: Behavioral: Reading Newspaper; Behavioral: Barlab-Exposure

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Test to induce high levels of acute social stress, including actors and a faked exam situation
  Arms: Social Stress Test
Behavioral: Reading Newspaper — Participants read newspaper
  Arms: Control Condition
Behavioral: Barlab-Exposure — Participants are exposed to a bar situation with different sorts of alcohol available. They sniff at water and at one alcoholic drink.

SUMMARY:
In this feasibility study the investigators are using a setup of stress-related body sensors including established as well as innovative sensor-based measures to identify predictor profiles for alcohol-related behavioral and neural measures in Alcohol Use Disorder (AUD). Long-term aim is the definition of a setup of mobile sensors and their integration in a mobile infrastructure that allows the prediction of stress related alcohol intake in an ambulatory setting.

DETAILED DESCRIPTION:
The long-term aim is the definition of a setup of mobile sensors and their integration in a mobile infrastructure that allows the prediction of stress related alcohol intake in an ambulatory setting.

In patients with Alcohol Use Disorder (AUD) stress exposure is known to affect craving, cue-reactivity and relapse risk. Here, the investigators aim to identify stress- and alcohol cue-related physiological markers in a lab experiment to assess interactions between acute psychological stress exposure and alcohol cue-exposure regarding their effects on alcohol craving and related markers (attentional bias to alcohol-cues, implicit association task, neural cue-reactivity). In addition to applying established stress-related markers (cortisol in saliva, heart-rate variability, systolic blood pressure and electrodermal activity), the investigators will integrate innovative measures currently under investigation (e.g. voice stress analysis) to identify whether these additional parameters increase the predictive significance.

ELIGIBILITY:
Inclusion Criteria:

* Heavy drinking, defined by alcohol consumption of at least 20g alcohol per day (at 5 days per week)
* sufficient ability to communicate with the investigators, to answer questions in oral and written form
* fully informed consent
* written informed consent

Exclusion Criteria:

* withdrawal of the declaration of consent
* positive urin drug screening (cannabis, amphetamine, opiates, benzodiazepines, cocaine)
* Lifetime history of DSM-5 bipolar disorder, schizophrenia or schizophrenia spectrum disorder, or substance dependence other than alcohol or nicotine or cannabis dependence.
* Current threshold DSM-5 diagnosis of major depressive disorder, or presence of suicidal intention
* History of severe head trauma or other severe central nervous system disorder (e.g., dementia, Parkinson's disease, multiple sclerosis)
* Current use of medications or drugs known to interact with the CNS within at least four half-lives post last intake

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
change in heart rate | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hours; starting 1 hour 50 minutes after arrival of the proband
  heart rate acquired with ear clip (continuous time series)
change in heart rate variability | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hours; starting 1 hour 50 minutes after arrival of the proband
  heart rate variability acquired with ear clip (continuous time series)
change in blood pressure (systolic and diastolic) | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at 2:20h, 2:50h, 3:20h, 3:50h, 4:50h, 5:05h after arrival of the proband
  acquired with pressure sleeve
change in electrodermal activity | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hour; starting 1h 50min after arrival of the proband
  time series acquired with body sensor
neural alcohol-related cue-reactivity | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; paradigm Vollstädt-Klein et al. 2010 [% signal change is not a change over time; it is measured during one experimental session]
neural inhibition processing | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; stop-signal reaction time task (Fauth-Buhler et al. 2012) [% signal change is not a change over time; it is measured during one experimental session]
neural emotion processing | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; faces task (Hariri et al. 2002) [% signal change is not a change over time; it is measured during one experimental session]
resting state activity | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  resting state connectivity measured with fMRI
attentional bias to alcohol cues | at examination day: measured directly after the stress task / newspaper reading; before "implicit alcohol association" and MRI session
  measured with reaction time differences (in milliseconds) using the dotprobe-task (Vollstädt-Klein et al. 2009) [reaction time differences is not a change over time; it is measured during one experimental session]
implicit alcohol association | at examination day: measured after the stress task / newspaper reading, directly after the "attentional bias to alcohol cues" ; before MRI session
  measured with reaction time differences (in milliseconds) using the implicit association task (Wiers et al. 2016) [reaction time differences is not a change over time; it is measured during one experimental session]
change in level of cortisol | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  cortisol measured in saliva as a stress marker
change in voice stress pattern | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  audio file of participants' voice for voice stress pattern analysis will be recorded. From this a multivariate measure (i.e. multivariate vector) will be acquired (including frequency, loudness etc.)
change in alcohol urges | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  elf-report questionnaire: "Alcohol Urge Questionnaire (AUQ)"; Bohn et al. 1995
change in alcohol craving | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  self-report "How strong is your craving for alcohol?": reported on a visual analogue scale ranging from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany